CLINICAL TRIAL: NCT06546345
Title: Effectiveness and Safety of the Silicone Joint Implant KeriFlex® and of Its Associated Instruments in the Treatment of MCP and PIP Arthritis: Post Market Clinical Follow up
Brief Title: Post Market Clinical Follow-Up KeriFlex®
Status: Recruiting | Type: Observational
Sponsor: Keri Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A01089-34
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis; Degenerative Arthritis; Traumatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: KeriFlex® — The KeriFlex® finger joint prothesis MCP is designed to replace a damaged metacarpophalangeal (MCP) joint and the KeriFlex® finger joint prothesis PIP is designed to replace a damaged proximal interphalangeal (PIP) joint.

SUMMARY:
The general objective of this study is to assess the performance and safety of the KeriFlex® silicone joint implant and its associated instruments, used in accordance with the labeling and instructions in force.

The performance and safety of the KeriFlex® joint implant will be established in the short and long term with regard to the life cycle of the implant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Patients who are going to undergo arthroplasty of the metacarpophalangeal or proximal interphalangeal joint using a KeriFlex® implant in accordance with the instructions for use and the labelling in force.
* Patients with rheumatoid arthritis, osteoarthritis or post-traumatic osteoarthritis

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with an intellectual disability who cannot follow their surgeon's instructions
* Patients with general surgery contraindications and particularly to the implantation of a KeriFlex® implant
* Patients with acute or chronic, local or systemic infections
* Metacarpal or phalanx destruction or poor bone quality preventing adequate fixation
* Muscle loss, alteration or vascular deficiency in the affected finger
* Patients with significant physical activity involving treated joint
* Children, young growing patients with open epiphyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any type of population requiring a surgical procedure covered by the device and presenting bone quality deemed satisfactory by the surgeon.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effectiveness of the KeriFlex® implant in improving the functional results of the hand | 6 months
  Proportion of patients with a bMHQ score greater than the preoperative value at 6 months (postoperative).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Jean Minjoz, Besançon
  - Clinic Lille Sud, Lesquin
  - Institut aquitain de la main et du membre supérieur, Pessac